CLINICAL TRIAL: NCT02939183
Title: (INTREPID-1) A Phase 1b Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of Oprozomib in Combination With Pomalidomide and Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Phase 1b Study Evaluating OPomD in Relapsed or Refractory Multiple Myeloma
Acronym: INTREPID-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20160104
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Dosage Forms; Dexamethasone; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1 Oprozomib Immediate-release (IR) + Dexamethasone (Experimental): Oprozomib IR plus dexamethasone
  Interventions: Drug: Immediate Release (IR) Formulation; Drug: Dexamethasone
- Part 1 Oprozomib Gastro-retentive (GR) + Dexamethasone (Experimental): Oprozomib GR plus dexamethasone
  Interventions: Drug: Gastro-Retentive (GR) Formulation; Drug: Dexamethasone
- Part 2 Oprozomib IR + Pomalidomide + Dexamethasone (Experimental): Oprozomib IR plus pomalidomide and dexamethasone
  Interventions: Drug: Immediate Release (IR) Formulation; Drug: Dexamethasone; Drug: Pomalidomide
- Part 2 Oprozomib GR + Pomalidomide + Dexamethasone (Experimental): Oprozomib GR plus pomalidomide and dexamethasone
  Interventions: Drug: Gastro-Retentive (GR) Formulation; Drug: Dexamethasone; Drug: Pomalidomide
- Open-label Roll-over (Experimental): Oprozomib GR monotherapy, or oprozomib GR plus dexamethasone
  Interventions: Drug: Gastro-Retentive (GR) Formulation; Drug: Dexamethasone

INTERVENTIONS:
Drug: Immediate Release (IR) Formulation — Immediate Release (IR) Formulation
  Arms: Part 1 Oprozomib Immediate-release (IR) + Dexamethasone; Part 2 Oprozomib IR + Pomalidomide + Dexamethasone
Drug: Gastro-Retentive (GR) Formulation — Gastro-Retentive (GR) Formulation
  Arms: Open-label Roll-over; Part 1 Oprozomib Gastro-retentive (GR) + Dexamethasone; Part 2 Oprozomib GR + Pomalidomide + Dexamethasone
Drug: Dexamethasone — Dexamethasone
Drug: Pomalidomide — Pomalidomide
  Arms: Part 2 Oprozomib GR + Pomalidomide + Dexamethasone; Part 2 Oprozomib IR + Pomalidomide + Dexamethasone

SUMMARY:
A study evaluating two new formulations of oprozomib plus pomalidomide and dexamethasone in participants with relapsed refractory multiple myeloma.

DETAILED DESCRIPTION:
A multicenter, non-randomized, open-label, dose-exploration study evaluating two new formulations of oprozomib plus pomalidomide and dexamethasone in participants with relapsed refractory multiple myeloma. The study will be conducted in two parts. Part 1 will evaluate the formulations of oprozomib in combination with dexamethasone only. Part 2 will evaluate the formulations of oprozomib administered at increasing dose levels (dose escalation) in combination with pomalidomide and dexamethasone.

ELIGIBILITY:
Inclusion criteria

* Participant must have a pathologically documented, definitively diagnosed, multiple myeloma relapse, or refractory progressive disease after at least 2 lines of therapy for multiple myeloma. Prior therapeutic treatment or regimens must include a proteasome inhibitor and lenalidomide.
* Participant must be willing and able to undergo bone marrow aspirate per protocol (with or without bone marrow biopsy per institutional guidelines).
* Measurable disease (assessed within 28 days prior to day 1).
* Eastern Cooperative Oncology Group (ECOG) performance status of <= 2.
* Other Inclusion Criteria May Apply

Exclusion Criteria

* Currently receiving treatment in another investigational device or drug study, or less than 28 days or 5 half-lives whichever is shorter since ending treatment on another investigational device or drug study(s).
* Previously received an allogeneic stem cell transplant and the occurrence of one or more of the following: received the transplant within 6 months prior to study day 1; received immunosuppressive therapy within the last 3 months prior to study day 1; having signs or symptoms of acute or chronic graft-versus-host disease.
* Autologous stem cell transplant < 90 days prior to study day 1.
* Multiple myeloma with IgM subtype.
* POEM syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
* Plasma cell leukemia (> 2.0 X10^9/L circulating plasma cells by standard differential).
* Waldenstrom's macroglobulinemia.
* Other Exclusion Criteria May Apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (20):
- United States (13):
  - Research Site, West Hollywood, California
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Bethesda, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Hackensack, New Jersey
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, San Antonio, Texas
  - Research Site, Milwaukee, Wisconsin
- Australia (3):
  - Research Site, Clayton, Victoria
  - Research Site, Murdoch, Western Australia
  - Research Site, Perth, Western Australia
- Canada (2):
  - Research Site, Calgary, Alberta
  - Research Site, Toronto, Ontario
- Spain (2):
  - Research Site, Salamanca, Castille and León
  - Research Site, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 26 research centers in Australia, Canada, Spain, and the United States, and participated from 17 January 2017 to 06 October 2022.
Pre-assignment Details: Part 1 evaluated oprozomib formulations (immediate-release [IR] and gastro-retentive [GR]) administered at a 150 mg/day dose level with dexamethasone. Part 2 evaluated the IR and GR oprozomib formulations administered at different increasing dose levels with pomalidomide and dexamethasone. An open-label roll-over part was conducted in the United States to include eligible participants from separate Amgen oprozomib studies in a single arm as pre-specified in the statistical analysis plan (SAP).
Groups:
- Oprozomib IR 150 mg/Day + Dexamethsone: In Part 1, participants received oprozomib IR 150 mg/day administered orally every week on 2 consecutive days (2/7 schedule) in combination with dexamethasone 20 mg orally (days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle), for up to 10 months.
- Oprozomib GR 150 mg/Day + Dexamethasone: In Part 1, participants received oprozomib GR 150 mg/day administered orally every week on 2 consecutive days (2/7 schedule) in combination with dexamethasone 20 mg orally (days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle), for up to 10 months.
- Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone: In Part 2, participants received oprozomib IR 150 mg/day administered orally every week on 2 consecutive days (2/7 schedule) in combination with dexamethasone 20 mg orally (days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle), for up to 10 months. Participants also received pomalidomide 4 mg orally once daily on days 1 to 21 of each 28-day cycle.
- Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone: In Part 2, participants received oprozomib GR 150 mg/day administered orally every week on 2 consecutive days (2/7 schedule) in combination with dexamethasone 20 mg orally (days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle), for up to 10 months. Participants also received pomalidomide 4 mg orally once daily on days 1 to 21 of each 28-day cycle.
- Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone: In Part 2, participants received oprozomib IR 150 mg/day on days 1 and 2 of cycle 1, and oprozomib IR 200 mg/day administered orally every week on 2 consecutive days from cycle 1 day 8 onwards (2/7 schedule), for up to 10 months. Participants also received dexamethasone 20 mg orally (days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle), and pomalidomide 4 mg orally once daily on days 1 to 21 of each 28-day cycle.
- Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone: In Part 2, participants received oprozomib GR 150 mg/day on days 1 and 2 of cycle 1, and oprozomib GR 200 mg/day administered orally every week on 2 consecutive days from cycle 1 day 8 onwards (2/7 schedule), for up to 10 months. Participants also received dexamethasone 20 mg orally (days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle), and pomalidomide 4 mg orally once daily on days 1 to 21 of each 28-day cycle.
- Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone: In Part 2, participants received oprozomib IR 150 mg/day on days 1 and 2 of cycle 1, and oprozomib IR 225 mg/day administered orally every week on 2 consecutive days from cycle 1 day 8 onwards (2/7 schedule), for up to 10 months. Participants also received dexamethasone 20 mg orally (days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle), and pomalidomide 4 mg orally once daily on days 1 to 21 of each 28-day cycle.
- Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone: In Part 2, participants received oprozomib IR 150 mg/day on days 1 and 2 of cycle 1, and oprozomib IR 250 mg/day administered orally every week on 2 consecutive days from cycle 1 day 8 onwards (2/7 schedule), for up to 10 months. Participants also received dexamethasone 20 mg orally (days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle), and pomalidomide 4 mg orally once daily on days 1 to 21 of each 28-day cycle.
- Open-label Roll-over: Eligible participants who had enrolled on separate Amgen oprozomib studies (2011-001 [NCT01416428], 2012-001 [NCT01832727], OPZ003 [NCT01881789], OPZ007 [NCT01999335], and OPZ009 [NCT02244112]) and were receiving oprozomib as monotherapy, or a combination of oprozomib with dexamethasone, continued treatment in research centers within the United States only. Participants continued receiving the previous dose/schedule of oprozomib GR formulation until disease progression, death, or unacceptable toxicity.
Period: Overall Study
Arm/Group | Oprozomib IR 150 mg/Day + Dexamethsone | Oprozomib GR 150 mg/Day + Dexamethasone | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone | Open-label Roll-over
Started | 5 | 8 | 3 | 5 | 9 | 5 | 11 | 8 | 7
Received Oprozomib | 5 | 8 | 3 | 4 | 9 (1 participant enrolled in arm Oprozomib IR 200 mg/day + pomalidomide + dexamethasone received oprozomib IR 150 mg + pomalidomide + dexamethasone.) | 5 | 10 | 8 | 7
Completed | 5 | 5 | 2 | 2 | 7 | 3 | 4 | 5 | 1
Not Completed | 0 | 3 | 1 | 3 | 2 | 2 | 7 | 3 | 6
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Sponsor decision | 0 | 1 | 0 | 1 | 2 | 0 | 3 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 2 | 2
Not completed — Not treated due to adverse event | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received any amount of oprozomib, pomalidomide and/or dexamethasone. One participant in arm Oprozomib IR 200 mg/day + pomalidomide + dexamethasone received oprozomib IR 150 mg + pomalidomide + dexamethasone, and their baseline characteristics data were included in the Oprozomib IR 150 mg + pomalidomide + dexamethasone arm. Participants enrolled from other Amgen studies were included in a single roll-over arm, as pre-specified in the SAP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oprozomib IR 150 mg/Day + Dexamethsone | Oprozomib GR 150 mg/Day + Dexamethasone | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone | Open-label Roll-over | Total
Number analyzed (Participants) | 5 | 8 | 4 | 4 | 8 | 5 | 10 | 8 | 7 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (17.2) | 59.6 (8.1) | 62.5 (8.7) | 63.5 (5.9) | 64.3 (9.8) | 62.0 (8.2) | 63.1 (10.2) | 65.9 (10.5) | 70.4 (8.7) | 63.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 2 | 1 | 3 | 3 | 3 | 1 | 1 | 19
  Male | 4 | 4 | 2 | 3 | 5 | 2 | 7 | 7 | 6 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 8 | 4 | 4 | 8 | 5 | 7 | 8 | 7 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black (or African American) | 1 | 1 | 2 | 0 | 1 | 2 | 2 | 1 | 0 | 10
  White | 4 | 7 | 2 | 4 | 6 | 3 | 7 | 7 | 6 | 46
  Other | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxcity (DLT)
Description: DLTs were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 and included the below, if judged by the investigator/medical monitor to be possibly related to study treatment: Non-hematologic DLTs were any ≥ Grade 3 toxicity, except: Grade 3 asymptomatic electrolyte abnormalities (except hypophosphatemia > 24 hours); Grade 3 nausea, vomiting and diarrhea < 3 days; Grade 3 fatigue < 14 days; ≥ Grade 3 hyperglycemia/toxicity due to dexamethasone; ≥ Grade 3 rash due to pomalidomide. Hematologic DLTs included: Grade 4 neutropenia if absolute neutrophil count < 0.5 x 10^9/L ≥ 7 days; febrile neutropenia; Grade 4 thrombocytopenia ≥ 7 days; Grade ≥ 3 with ≥ Grade 2 bleeding/requiring platelet transfusion.
Time Frame: Day 1 to day 28 of cycle 1, where each cycle was 28 days
Population: DLT-evaluable participants received the following during the 28-day DLT window: all planned doses of oprozomib, a minimum of 17 of 21 planned doses of pomalidomide, and a minimum of 6 of 8 planned doses of dexamethasone. One participant enrolled in arm Oprozomib IR 200 mg/day + pomalidomide + dexamethasone received oprozomib IR 150 mg + pomalidomide + dexamethasone, and this participant was included in the Oprozomib IR 150 mg + pomalidomide + dexamethasone arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Oprozomib IR 150 mg/Day + Dexamethsone | Oprozomib GR 150 mg/Day + Dexamethasone | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 5 | 8 | 4 | 4 | 8 | 5 | 10 | 8
Participants | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Each Formulation of Oprozomib in Combination With Pomolidomide and Dexamethasone
Description: The MTD was the dose with the highest posterior probability of having a DLT rate within the target toxicity interval (15% to 25%), while the posterior probability of excessive/unacceptable toxicity (>25% to 100%) is <40%.
  DLTs were graded using CTCAE version 4.03 and included the below, if judged by the investigator/medical monitor to be possibly related to study treatment: Non-hematologic DLTs were any ≥ Grade 3 toxicity, except: Grade 3 asymptomatic electrolyte abnormalities (except hypophosphatemia > 24 hours); Grade 3 nausea, vomiting and diarrhea < 3 days; Grade 3 fatigue < 14 days; ≥ Grade 3 hyperglycemia/toxicity due to dexamethasone; ≥ Grade 3 rash due to pomalidomide. Hematologic DLTs included: Grade 4 neutropenia if absolute neutrophil count < 0.5 x 10^9/L ≥ 7 days; febrile neutropenia; Grade 4 thrombocytopenia ≥ 7 days; Grade ≥ 3 with ≥ Grade 2 bleeding/requiring platelet transfusion.
Time Frame: Day 1 to Day 28 of cycle 1, where each cycle was 28 days
Population: DLT-evaluable participants in Part 2 who received the following during the 28-day DLT window: all planned doses of oprozomib, a minimum of 17 of 21 planned doses of pomalidomide, and a minimum of 6 of 8 planned doses of dexamethasone.
Measure: Number; unit: mg/day
Groups:
- All Doses Oprozomib IR + Pomalidomide + Dexamethasone: Participants who received oprozomib IR in a 2/7 schedule in combination with pomalidomide and dexamethasone in Part 2. Doses of oprozomib IR administered were 150 mg/day (N=4), 200 mg/day (N=8), 225 mg/day (N=10), and 250 mg/day (N=8).
- All Doses Oprozomib GR + Pomalidomide + Dexamethasone: Participants who received oprozomib GR in a 2/7 schedule in combination with pomalidomide and dexamethasone in Part 2. Doses of oprozomib GR administered were 150 mg/day (N=4), and 200 mg/day (N=5).
Arm/Group | All Doses Oprozomib IR + Pomalidomide + Dexamethasone | All Doses Oprozomib GR + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 30 | 9
mg/day | 250 | NA — The MTD for oprozomib GR in combination with pomalidomide and dexamethasone was not determined due to too few DLTs.

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) (Oprozomib in Combination With Dexamethasone and/or Pomalidomide)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant. TEAEs were any AE that started on or after receiving the first dose of investigational product and up to and including 30 days after the last dose of investigational product or the end of study date, whichever is earlier. Treatment-related TEAEs were those considered related to study treatment by the investigator. Any clinically significant changes in electrocardiograms, vital signs, physical examination with a neurological assessment and clinical laboratory tests were recorded as TEAEs.
Time Frame: Day 1 of cycle 1 to 30 (+7) days after the last dose of study treatment or end of study date, whichever is earlier (where each cycle was 28 days). Median treatment duration in Part 1 was 11.43 weeks and in Part 2 was 28 weeks
Population: Participants in the safety analysis set who received any amount of oprozomib, pomalidomide and/or dexamethasone in Parts 1 and 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Oprozomib IR 150 mg/Day + Dexamethsone | Oprozomib GR 150 mg/Day + Dexamethasone | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 5 | 8 | 4 | 4 | 8 | 5 | 10 | 8
Participants
  Any TEAE | 4 | 8 | 4 | 4 | 8 | 5 | 10 | 8
  Any Treatment-related TEAE | 4 | 8 | 4 | 4 | 8 | 5 | 10 | 8

4. Primary Outcome: Number of Participants With TEAEs and Treatment-emergent Serious AEs (Open-label Roll-over)
Description: TEAEs were any AE that started on or after receiving the first dose of investigational product and up to and including 30 days after the last dose of investigational product or the end of study date, whichever is earlier. Treatment-related TEAEs were those considered related to study treatment by the investigator. Serious TEAEs were any AE meeting at least 1 of the following criteria: fatal; life-threatening; required in-patient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; congenital anomaly/birth defect; other medically important serious event.
Time Frame: Day 1 to 30 (+7) days after the last dose of study treatment or end of study date, whichever is earlier (where each cycle was 28 days). Median treatment duration for the open-label roll-over arm was 75.14 weeks
Population: The safety analysis set for roll-over participants included all roll-over participants who received any amount of oprozomib, pomalidomide and/or dexamethasone. Participants enrolled in this study from other Amgen studies were included in a single roll-over arm, as pre-specified in the SAP.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Roll-over
Number analyzed (Participants) | 7
Participants
  Any TEAE | 7
  Any Serious TEAE | 4

5. Secondary Outcome: Maximum Observed Concentration (Cmax) of Oprozomib
Description: The mean Cmax of oprozomib is presented following dosing on cycle 1 day 8 and cycle 1 day 22 for the IR and GR oprozomib formulations.
Time Frame: Cycle 1 days 8 and 22: pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose. GR only: cycle 1 day 8: 8 hours post-dose
Population: Participants in the PK analysis set with data available at each time point. The PK analysis set included participants for whom at least 1 PK parameter could be adequately estimated, excluding roll-over participants.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oprozomib IR 150 mg/Day + Dexamethsone | Oprozomib GR 150 mg/Day + Dexamethasone | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 7 | 5 | 10 | 7
ng/mL
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 3 | 3 | 7 | 5 | 10 | 7
  Cycle 1 Day 8 | 321 (89.2) | 118 (90.3) | 349 (195) | 119 (77.7) | 694 (479) | 367 (429) | 1020 (911) | 800 (703)
  Cycle 1 Day 22: number analyzed (Participants) | 3 | 6 | 1 | 3 | 4 | 4 | 10 | 4
  Cycle 1 Day 22 | 453 (48.0) | 209 (185) | 305 (NA) — Standard deviation (SD) could not be determined due to too few participants with available data at this time point. | 191 (99.2) | 1040 (941) | 137 (81.1) | 1580 (672) | 1420 (1250)

6. Secondary Outcome: Time to Cmax (Tmax) of Oprozomib
Description: The median Tmax of oprozomib is presented following dosing on cycle 1 day 8 and cycle 1 day 22 for the IR and GR oprozomib formulations.
Time Frame: Cycle 1 days 8 and 22: pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose. GR only: cycle 1 day 8: 8 hours post-dose
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Oprozomib IR 150 mg/Day + Dexamethsone | Oprozomib GR 150 mg/Day + Dexamethasone | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 7 | 5 | 10 | 7
hours
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 3 | 3 | 7 | 5 | 10 | 7
  Cycle 1 Day 8 | 1.0 [0.93 to 1.9] | 2.0 [2.0 to 4.0] | 2.0 [0.50 to 2.0] | 5.8 [3.9 to 6.0] | 2.0 [0.45 to 6.0] | 2.0 [1.1 to 5.8] | 1.5 [0.47 to 4.2] | 1.3 [0.42 to 5.8]
  Cycle 1 Day 22: number analyzed (Participants) | 3 | 6 | 1 | 3 | 4 | 4 | 10 | 4
  Cycle 1 Day 22 | 1.0 [0.98 to 2.0] | 3.0 [1.9 to 6.0] | 1.0 [1.0 to 1.0] | 4.1 [3.7 to 6.0] | 1.3 [0.45 to 2.0] | 4.8 [2.0 to 6.0] | 0.98 [0.42 to 2.2] | 0.75 [0.50 to 1.1]

7. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Oprozomib
Description: The mean AUClast of oprozomib is presented following dosing on cycle 1 day 8 and cycle 1 day 22 for the IR and GR oprozomib formulations.
Time Frame: Cycle 1 days 8 and 22: pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose. GR only: cycle 1 day 8: 8 hours post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Oprozomib IR 150 mg/Day + Dexamethsone | Oprozomib GR 150 mg/Day + Dexamethasone | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 7 | 5 | 10 | 7
hour*ng/mL
  Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 3 | 3 | 7 | 5 | 10 | 7
  Cycle 1 Day 8 | 656 (77.6) | 357 (252) | 869 (449) | 655 (73.5) | 1210 (658) | 1880 (2190) | 1730 (1160) | 1710 (1560)
  Cycle 1 Day 22: number analyzed (Participants) | 3 | 6 | 1 | 3 | 4 | 4 | 10 | 4
  Cycle 1 Day 22 | 1020 (281) | 1380 (1090) | 681 (NA) — The SD could not be determined due to too few participants with available data at this time point. | 839 (544) | 1420 (659) | 888 (1200) | 2050 (722) | 2030 (1070)

8. Secondary Outcome: Best Overall Response (BOR) According to Revised International Myeloma Working Group Uniform Response Criteria (IMWG-URC)
Description: BOR was the best response per IMWG-URC from best to worst: stringent complete response (sCR; complete response [CR], normal serum free light chain ratio, no clonal cells in bone marrow [BM]), CR (negative immunofixation on serum and urine, soft tissue plasmacytomas disappearance, < 5% plasma cells in BM), very good partial response (VGPR; serum and urine M-protein detectable by immunofixation or ≥ 90% reduction in serum M-protein [urine M-protein level < 100 mg/24-h]), partial response (PR; ≥ 50% reduction of serum M-protein and 24-h urinary M-protein by ≥ 90% or < 200 mg/24-h), minimal response (MR; 25-49% reduction of serum M-protein and 50-89% in 24-h urinary M-protein, exceeding 200 mg/24-h), stable disease (SD; not CR, VGPR, PR or progressive disease [PD]), and PD (≥ 25% increase in serum or urine M-component, development of new or increased size of existing bone lesions or soft tissue plasmacytomas, hypercalcemia attributed to the plasma cell proliferative disorder).
Time Frame: Day 1 of cycle 1 up to the end of study visit (where each cycle was 28 days); median treatment duration in Part 1 was 11.43 weeks and in Part 2 was 28 weeks
Population: The efficacy analysis set included all participants, excluding roll-over participants, who were included in the safety analysis set, and had a baseline disease assessment and at least 1 post-baseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Oprozomib IR 150 mg/Day + Dexamethsone | Oprozomib GR 150 mg/Day + Dexamethasone | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 7 | 5 | 10 | 8
Participants
  sCR | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  VGPR | 1 | 0 | 0 | 0 | 3 | 0 | 2 | 3
  PR | 1 | 1 | 1 | 0 | 3 | 2 | 3 | 3
  MR | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
  SD | 0 | 4 | 0 | 1 | 0 | 0 | 4 | 0
  PD | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unconfirmed response | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 1

9. Secondary Outcome: Overall Response Rate (ORR) According to IMWG-URC
Description: The ORR was defined as the percentage of participants with a BOR of sCR, CR, VGPR, and PR per the IMWG-URC. Complete response (CR): Negative immunofixation on serum and urine, soft tissue plasmacytomas disappearance, < 5% plasma cells in bone marrow (BM). Stringent CR (sCR): CR and normal serum free light chain ratio and no clonal cells in BM. Very Good Partial Response (VGPR): Serum and urine M-protein detectable by immunofixation or ≥ 90% reduction in serum M-protein (urine M-protein level < 100 mg/24-h). PR: ≥ 50% reduction of serum M-protein and 24-h urinary M-protein by ≥ 90% or to < 200 mg/24-h. The 95% confidence intervals (CIs) were estimated using the Clopper-Pearson method.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oprozomib IR 150 mg/Day + Dexamethsone | Oprozomib GR 150 mg/Day + Dexamethasone | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 7 | 5 | 10 | 8
percentage of participants | 66.7 [9.4 to 99.2] | 16.7 [0.4 to 64.1] | 33.3 [0.8 to 90.6] | 0.0 [NA to NA] — The 95% CIs could not be determined as no participants achieved OR. | 85.7 [42.1 to 99.6] | 60.0 [14.7 to 94.7] | 60.0 [26.2 to 87.8] | 87.5 [47.3 to 99.7]

10. Secondary Outcome: Number of Participants With Progression Free Survival (PFS) Events
Description: PFS was defined as the number of months from a participant's first dose of study treatment to the earlier of disease progression or death due to any cause. The number of participants who had a PFS event or who were censored are presented. PFS events were an assessment of progressive disease according to the IMWG-URC or death due to any cause. PFS data was censored: participants alive and no documented disease progression at time of analysis were censored at date of last disease assessment; participants alive with no disease assessment were censored at the first study dose date; participants alive without documented disease progression, with withdrawn consent were censored at date of last disease assessment before consent withdrawal; and for participants who started anti-cancer therapy other than study treatment prior to documentation of disease progression were censored at date of last disease assessment prior to starting new therapy.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Oprozomib IR 150 mg/Day + Dexamethsone | Oprozomib GR 150 mg/Day + Dexamethasone | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 7 | 5 | 10 | 8
Participants
  Participants with PFS events | 0 | 1 | 1 | 0 | 0 | 2 | 4 | 1
  Participants who were censored | 3 | 5 | 2 | 3 | 7 | 3 | 6 | 7

11. Secondary Outcome: Kaplan-Meier Estimate of PFS
Description: PFS was defined as the number of months from a participant's first dose of study treatment to the earlier of disease progression or death due to any cause. Median PFS was estimated using the Kaplan-Meier method. 95% CIs were estimated using the method by Klein and Moeschberger (1997) with log-log transformation. PFS data was censored: participants alive and no documented disease progression at time of analysis were censored at date of last disease assessment; participants alive with no disease assessment were censored at the first study dose date; participants alive without documented disease progression, with withdrawn consent were censored at date of last disease assessment before consent withdrawal; and for participants who started anti-cancer therapy other than study treatment prior to documentation of disease progression were censored at date of last disease assessment prior to starting new therapy.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oprozomib IR 150 mg/Day + Dexamethsone | Oprozomib GR 150 mg/Day + Dexamethasone | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 7 | 5 | 10 | 8
months | NA [NA to NA] — The median and upper and lower 95% CIs could not be estimated due to too few events. | NA [2.7 to NA] — The median and upper 95% CI could not be estimated due to too few events. | 14.24 [NA to NA] — Due to the low numbers of participants (3) there are too few events (1) that impacted the estimate of survival function to no variation, hence the 95% CIs could not be estimated. | NA [NA to NA] — The median and upper and lower 95% CIs could not be estimated due to too few events. | NA [NA to NA] — The median and upper and lower 95% CIs could not be estimated due to too few events. | NA [1.5 to NA] — The median and upper 95% CI could not be estimated due to too few events. | 17.50 [5.6 to NA] — The upper 95% CI could not be estimated due to too few events. | NA [29.5 to NA] — The median and upper 95% CI could not be estimated due to too few events.

12. Secondary Outcome: Kaplan-Meier Estimate of Duration of Response (DOR)
Description: DOR, presented in months, was defined as the number of days between the date of the first tumor assessment indicating an objective response (PR or better) through to the subsequent date of progression or death due to any cause, or where applicable date of censoring (date of first progressive disease assessment or death or date of censoring - date of the first objective response result + 1/30.4). Median PFS was estimated using the Kaplan-Meier method. 95% confidence intervals were estimated using the method by Klein and Moeschberger (1997) with log-log transformation.
Time Frame: as for outcome 8
Population: The efficacy analysis set included all participants, excluding roll-over participants, who were included in the safety analysis set, and had a baseline disease assessment and at least 1 post-baseline disease assessment. Participants who did not achieve an objective response were excluded from the analysis of DOR. Participants who responded and had not progressed while on study were censored at the date of assessment of the last evaluable tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oprozomib IR 150 mg/Day + Dexamethsone | Oprozomib GR 150 mg/Day + Dexamethasone | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone
Number analyzed (Participants) | 2 | 1 | 1 | 0 | 6 | 3 | 6 | 7
months | NA [NA to NA] — The median, upper and lower 95% CIs could not be estimated due to too few events. | NA [NA to NA] — The median, upper and lower 95% CIs could not be estimated due to too few events. | NA [NA to NA] — The median, upper and lower 95% CIs could not be estimated due to too few events. |  | NA [NA to NA] — The median, upper and lower 95% CIs could not be estimated due to too few events. | NA [NA to NA] — The median, upper and lower 95% CIs could not be estimated due to too few events. | 16.6 [3.7 to NA] — The upper 95% CI could not be estimated due to too few events. | NA [28.6 to NA] — The median could not be estimated due to too few events. The lower bound 95% CI was estimated from observed data that were available (25% percentile).

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the first dose of study treatment until the last dose + 30 days; median treatment duration in Part 1 was 11.43 weeks, in Part 2 was 28 weeks, and in the open-label roll-over arm was 75.14 weeks. All-cause mortality was collected from enrollment to end of study visit; median overall duration on study was 259.00 days.
Description: Serious adverse events and other adverse events are reported for all participants who received any amount of oprozomib, pomalidomide and/or dexamethasone (safety analysis set) and were collected according to treatment received. All-cause mortality is reported for all participants enrolled in the study and was collected according to assigned treatment group. Participants enrolled in this study from other Amgen studies were included in a single roll-over arm, as pre-specified in the SAP.
Arm/Group | Oprozomib IR 150 mg/Day + Dexamethsone | Oprozomib GR 150 mg/Day + Dexamethasone | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone | Open-label Roll-over
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/8 | 1/3 | 0/5 | 0/9 | 2/5 | 1/11 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/8 | 2/4 | 4/4 | 6/8 | 5/5 | 3/10 | 4/8 | 4/7
Other Adverse Events (participants affected / at risk) | 4/5 | 8/8 | 4/4 | 4/4 | 8/8 | 5/5 | 10/10 | 8/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oprozomib IR 150 mg/Day + Dexamethsone (N=5) | Oprozomib GR 150 mg/Day + Dexamethasone (N=8) | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone (N=4) | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone (N=4) | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone (N=8) | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone (N=5) | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone (N=10) | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone (N=8) | Open-label Roll-over (N=7)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pasteurella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 3 | 1 | 2 | 1 | 2 | 1
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stroke in evolution (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oprozomib IR 150 mg/Day + Dexamethsone (N=5) | Oprozomib GR 150 mg/Day + Dexamethasone (N=8) | Oprozomib IR 150 mg/Day + Pomalidomide + Dexamethasone (N=4) | Oprozomib GR 150 mg/Day + Pomalidomide + Dexamethasone (N=4) | Oprozomib IR 200 mg/Day + Pomalidomide + Dexamethasone (N=8) | Oprozomib GR 200 mg/Day + Pomalidomide + Dexamethasone (N=5) | Oprozomib IR 225 mg/Day + Pomalidomide + Dexamethasone (N=10) | Oprozomib IR 250 mg/Day + Pomalidomide + Dexamethasone (N=8) | Open-label Roll-over (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 3 | 1 | 2 | 2 | 3 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 2 | 1 | 3 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Steroid withdrawal syndrome (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Cataract nuclear (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctival disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 3 | 1 | 2 | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 3 | 2 | 1 | 4 | 3 | 3 | 6 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 3 | 2 | 5 | 4 | 8 | 8 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 7 | 3 | 3 | 6 | 3 | 8 | 8 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 2 | 1 | 6 | 3 | 7 | 7 | 1
Asthenia (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Catheter site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Chills (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 4 | 2 | 3 | 3 | 2 | 6 | 5 | 0
Feeling jittery (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 2 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 1 | 3 | 3 | 5 | 1 | 0
Pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 2 | 2 | 1 | 2 | 3 | 1
Secretion discharge (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Temperature regulation disorder (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Immunisation reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Moraxella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1 | 0 | 3 | 2 | 1 | 5 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 3 | 0 | 2 | 3 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Radiation injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Crystal urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 3 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Norovirus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 2 | 2 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 3 | 3 | 0 | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 3 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 3 | 3 | 2 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Headache (Nervous system disorders) | 0 | 3 | 0 | 0 | 1 | 2 | 2 | 4 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0
Intention tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasticity (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 1 | 0 | 2 | 1 | 6 | 3 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myeloma cast nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 2 | 2 | 2 | 5 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 1 | 2 | 2 | 4 | 3 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 0 | 1
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion removal (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT02939183/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT02939183/SAP_001.pdf